CLINICAL TRIAL: NCT00135707
Title: A Randomized Clinical Trial of Antioxidants to Prevent Preeclampsia and An Observational Cohort Study to Predict Preeclampsia
Brief Title: Combined Antioxidant and Preeclampsia Prediction Studies (CAPPS)
Acronym: CAPPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HD36801-CAPPS; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD027860 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U01HD036801 (NIH); U10HD053097 (NIH); U10HD053118 (NIH)
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Preeclampsia
Keywords: Antioxidants; Preeclampsia; Pregnancy; Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Dietary Supplements; Vitamins; Ascorbic Acid; alpha-Tocopherol; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Supplement/Vitamins (Experimental): 1000mg of Vitamin C and 400IU of Vitamin E per capsule, twice daily between randomization (at 9 to 16 weeks) up to delivery.
  Interventions: Drug: Dietary Supplement/Vitamins
- Placebo for Vitamin C and Vitamin E (Placebo Comparator): Placebo capsules consisting of Mineral Oil, Hydrogenated Vegetable Oil, Lecithin, Yellow wax, Soft Gelatin Shell, twice daily between randomization (at 9 to 16 weks) up to delivery.
  Interventions: Drug: Placebo for Vitamin C and Vitamin E

INTERVENTIONS:
Drug: Dietary Supplement/Vitamins — Vitamin C (1000 mg) and Vitamin E (400 IU) per capsule, two capsules daily between randomization (at 9 - 16 weeks gestation) up to delivery.
  Other Names: Ascorbic Acid and d-alpha-Tocopheryl Acetate
  Arms: Dietary Supplement/Vitamins
Drug: Placebo for Vitamin C and Vitamin E — Placebo two capsules daily between randomization (at 9 - 16 weeks gestation) up to delivery.
  Arms: Placebo for Vitamin C and Vitamin E

SUMMARY:
Preeclampsia is one of the most common complications of pregnancy and is characterized by high blood pressure and protein in the urine. This can cause problems in the second half of pregnancy for both the mother and fetus. This study of preeclampsia consists of two parts: 1) a randomized, placebo controlled, multicenter clinical trial of 10,000 low-risk nulliparous women between 9 and 16 weeks gestation and 2) an observational, cohort study of 4,000 patients between 9 and 12 weeks gestation who are also enrolled in the trial.

Subjects in both parts will receive either 1000 mg of vitamin C and 400 IU of vitamin E or matching placebo daily. The purpose of the randomized, clinical trial is to find out if high doses of vitamin C and E will reduce the risk of preeclampsia and other problems associated with the disease. The study will also evaluate the safety of antioxidant therapy for mother and infant. Patients will be seen monthly to receive their supply of study drug, to have weight and blood pressure recorded, to have urine protein measured, and to assess any side effects. At two visits, blood and urine will be collected.

The observational, cohort study will prospectively measure potential biochemical and biophysical markers that might predict preeclampsia. These patients will have additional procedures including uterine artery Doppler and blood drawn for a complete blood count (CBC).

DETAILED DESCRIPTION:
A Randomized, Clinical Trial of Antioxidants to Prevent Preeclampsia:

Preeclampsia is the leading cause of maternal morbidity, as well as perinatal morbidity and mortality. Once the diagnosis has been established, therapy other than delivery has not been successful except to prolong pregnancy minimally (at some risk to mother and infant). Prevention efforts to reduce or eliminate preeclampsia are directed at the pathophysiology of the disorder prior to clinically evident preeclampsia and before irreversible changes have occurred.

This double-masked, placebo-controlled trial of 10,000 subjects is designed to evaluate the effects of antioxidant therapy in preventing serious complications associated with pregnancy-related hypertension in low risk, nulliparous women who begin treatment at 9-16 weeks gestation. The hypothesis being tested is that antioxidant therapy initiated prior to 16 weeks gestation will reduce the frequency of serious maternal and infant complications associated with pregnancy-related hypertension.

After randomization, subjects will receive either 1000 mg of vitamin C and 400 IU of vitamin E or matching placebo daily. They will be seen for monthly pill counts and to assess side effects, weight, blood pressure, and urine for protein. Blood and urine are collected at 24 and 32 weeks' gestation.

An Observational Cohort Study to Predict Preeclampsia:

A prospective, cohort study has been designed to complement the randomized, controlled, trial (RCT) and will test various biochemical and biophysical markers for ability to predict preeclampsia in 4,000 of the women who are enrolled in the RCT and are between 9 and 12 weeks gestation. These subjects will have additional procedures including a CBC and uterine artery Doppler.

ELIGIBILITY:
RCT Inclusion Criteria:

* Gestational age 9 -16 weeks
* Singleton pregnancy
* Nulliparous

Observational Inclusion Criteria:

* Women randomized to the RCT
* Gestational age 9 - 12 wks

Exclusion Criteria RCT and Observational:

* BP >= 135/85
* Proteinuria
* History or current use of anti-hypertensive medication or diuretics
* Use of vitamins C > 150 mg and/or E > 75 IU per day
* Pregestational diabetes
* Current pregnancy is a result of in vitro fertilization
* Regular use of platelet active drugs or non-steroidal anti-inflammatory drugs (NSAIDS)
* Known fetal abnormalities
* Documented uterine bleeding within a week of screening
* Uterine malformations
* History of medical complications
* Illicit drug or alcohol abuse during current pregnancy
* Intent to deliver elsewhere
* Participating in another interventional study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10154 (Actual)
Dates: Start 2003-06; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Miodovnik, MD, Study Director — NICHD Project Scientist; Rebecca Clifton, Ph.D., Principal Investigator — George Washington University Biostatistics Center; James M Roberts, MD, Study Chair — University of Pittsburgh - Magee Womens
Locations (16):
- United States (16):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwest, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after completion of the trial an publication of the main analyses per NIH Policy. Requests should be emailed to mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Background] Hauth JC, Clifton RG, Roberts JM, Myatt L, Spong CY, Leveno KJ, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal insulin resistance and preeclampsia. Am J Obstet Gynecol. 2011 Apr;204(4):327.e1-6. doi: 10.1016/j.ajog.2011.02.024. PMID 21458622
- [Background] Carreno CA, Clifton RG, Hauth JC, Myatt L, Roberts JM, Spong CY, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Sciscione A, Tolosa JE, Saade GR, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Excessive early gestational weight gain and risk of gestational diabetes mellitus in nulliparous women. Obstet Gynecol. 2012 Jun;119(6):1227-33. doi: 10.1097/AOG.0b013e318256cf1a. Erratum In: Obstet Gynecol. 2012 Sep;120(3):710. Saade, George R [added]. PMID 22617588
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Hauth JC, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Iams JD, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. First-trimester prediction of preeclampsia in nulliparous women at low risk. Obstet Gynecol. 2012 Jun;119(6):1234-42. doi: 10.1097/AOG.0b013e3182571669. PMID 22617589
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Hauth JC, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Grobman WA, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). The utility of uterine artery Doppler velocimetry in prediction of preeclampsia in a low-risk population. Obstet Gynecol. 2012 Oct;120(4):815-22. doi: 10.1097/AOG.0b013e31826af7fb. PMID 22996099
- [Background] Weissgerber TL, Gandley RE, McGee PL, Spong CY, Myatt L, Leveno KJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Haptoglobin phenotype, preeclampsia risk and the efficacy of vitamin C and E supplementation to prevent preeclampsia in a racially diverse population. PLoS One. 2013;8(4):e60479. doi: 10.1371/journal.pone.0060479. Epub 2013 Apr 3. PMID 23573260
- [Background] Johnson J, Clifton RG, Roberts JM, Myatt L, Hauth JC, Spong CY, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Samuels P, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Pregnancy outcomes with weight gain above or below the 2009 Institute of Medicine guidelines. Obstet Gynecol. 2013 May;121(5):969-975. doi: 10.1097/AOG.0b013e31828aea03. PMID 23635732
- [Background] Myatt L, Clifton RG, Roberts JM, Spong CY, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Sciscione A, Tolosa JE, Saade G, Sorokin Y, Anderson GD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Can changes in angiogenic biomarkers between the first and second trimesters of pregnancy predict development of pre-eclampsia in a low-risk nulliparous patient population? BJOG. 2013 Sep;120(10):1183-91. doi: 10.1111/1471-0528.12128. Epub 2013 Jan 18. PMID 23331974
- [Background] Makhlouf MA, Clifton RG, Roberts JM, Myatt L, Hauth JC, Leveno KJ, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Iams JD, Sciscione A, Tolosa JE, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health Human Development Maternal-Fetal Medicine Units Network. Adverse pregnancy outcomes among women with prior spontaneous or induced abortions. Am J Perinatol. 2014 Oct;31(9):765-72. doi: 10.1055/s-0033-1358771. Epub 2013 Dec 17. PMID 24347257
- [Background] Cantu J, Clifton RG, Roberts JM, Leveno KJ, Myatt L, Reddy UM, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Samuels P, Sciscione A, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Laboratory abnormalities in pregnancy-associated hypertension: frequency and association with pregnancy outcomes. Obstet Gynecol. 2014 Nov;124(5):933-940. doi: 10.1097/AOG.0000000000000509. PMID 25437721
- [Background] Weissgerber TL, McGee PL, Myatt L, Hauth JC, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Samuels P, Sciscione AC, Harper M, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Haptoglobin phenotype and abnormal uterine artery Doppler in a racially diverse cohort. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1728-33. doi: 10.3109/14767058.2013.876622. Epub 2014 Jan 13. PMID 24345080
- [Background] Abramovici A, Gandley RE, Clifton RG, Leveno KJ, Myatt L, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman AM, Samuels P, Sciscione A, Harper M, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health Human Development Maternal-Fetal Medicine Units Network. Prenatal vitamin C and E supplementation in smokers is associated with reduced placental abruption and preterm birth: a secondary analysis. BJOG. 2015 Dec;122(13):1740-7. doi: 10.1111/1471-0528.13201. Epub 2014 Dec 17. PMID 25516497
- [Background] Basraon SK, Mele L, Myatt L, Roberts JM, Hauth JC, Leveno KJ, Varner MW, Wapner RJ, Thorp JM Jr, Peaceman AM, Ramin SM, Sciscione A, Tolosa JE, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Relationship of Early Pregnancy Waist-to-Hip Ratio versus Body Mass Index with Gestational Diabetes Mellitus and Insulin Resistance. Am J Perinatol. 2016 Jan;33(1):114-21. doi: 10.1055/s-0035-1562928. Epub 2015 Sep 9. PMID 26352680
- [Background] McDonnold M, Mele LM, Myatt L, Hauth JC, Leveno KJ, Reddy UM, Mercer BM; Eunice Kennedy Shriver National Institute of Child Health Human Development Maternal-Fetal Medicine Units (MFMU) Network. Waist-to-Hip Ratio versus Body Mass Index as Predictor of Obesity-Related Pregnancy Outcomes. Am J Perinatol. 2016 May;33(6):618-24. doi: 10.1055/s-0035-1569986. Epub 2016 Jan 20. PMID 26788786
- [Background] Hughes BL, Clifton RG, Hauth JC, Leveno KJ, Myatt L, Reddy UM, Varner MW, Wapner RJ, Mercer BM, Peaceman AM, Ramin SM, Tolosa JE, Saade G, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Is Mid-trimester Insulin Resistance Predictive of Subsequent Puerperal Infection? A Secondary Analysis of Randomized Trial Data. Am J Perinatol. 2016 Aug;33(10):983-90. doi: 10.1055/s-0036-1583188. Epub 2016 Apr 27. PMID 27120478
- [Background] Silver RM, Myatt L, Hauth JC, Leveno KJ, Peaceman AM, Ramin SM, Samuels P, Saade G, Sorokin Y, Clifton RG, Reddy UM. Cell-Free Total and Fetal DNA in First Trimester Maternal Serum and Subsequent Development of Preeclampsia. Am J Perinatol. 2017 Jan;34(2):191-198. doi: 10.1055/s-0035-1570383. Epub 2016 Jul 11. PMID 27398706
- [Background] Tita AT, Doherty L, Roberts JM, Myatt L, Leveno KJ, Varner MW, Wapner RJ, Thorp JM Jr, Mercer BM, Peaceman A, Ramin SM, Carpenter MW, Iams J, Sciscione A, Harper M, Tolosa JE, Saade GR, Sorokin Y; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Adverse Maternal and Neonatal Outcomes in Indicated Compared with Spontaneous Preterm Birth in Healthy Nulliparas: A Secondary Analysis of a Randomized Trial. Am J Perinatol. 2018 Jun;35(7):624-631. doi: 10.1055/s-0037-1608787. Epub 2017 Nov 30. PMID 29190847
- [Result] Roberts JM, Myatt L, Spong CY, Thom EA, Hauth JC, Leveno KJ, Pearson GD, Wapner RJ, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Carpenter MW, Samuels P, Sciscione A, Harper M, Smith WJ, Saade G, Sorokin Y, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Vitamins C and E to prevent complications of pregnancy-associated hypertension. N Engl J Med. 2010 Apr 8;362(14):1282-91. doi: 10.1056/NEJMoa0908056. PMID 20375405
- [Result] Hauth JC, Clifton RG, Roberts JM, Spong CY, Myatt L, Leveno KJ, Pearson GD, Varner MW, Thorp JM Jr, Mercer BM, Peaceman AM, Ramin SM, Sciscione A, Harper M, Tolosa JE, Saade G, Sorokin Y, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Vitamin C and E supplementation to prevent spontaneous preterm birth: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):653-658. doi: 10.1097/AOG.0b013e3181ed721d. PMID 20733448
- See also: The public website of the NICHD Maternal-Fetal Medicine Units (MFMU) Network — http://www.bsc.gwu.edu/mfmu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted from July 2003 through February 2008 at the 16 clinical centers and the independent data coordinating center of the MFMU Network. Gestational age at randomization was between 9 weeks 0 days and 16 weeks 6 days. Women were eligible for inclusion if they had not had a previous pregnancy that lasted beyond 19 weeks 6 days.
Pre-assignment Details: Women who were no more than 15 weeks pregnant and who consented to participate in the study were given a supply of placebo and asked to return within 2 weeks. Those who returned, who had taken at least 50% of the placebo they were supposed to have taken, and who still met the eligibility criteria were randomly assigned to receive study drug.
Groups:
- Vitamins: Vitamins C & E
- Placebo: Mineral Oil, Hydrogenated Vegetable Oil, Lecithin, Yellow wax, Soft Gelatin Shell
Period: Overall Study
Arm/Group | Vitamins | Placebo
Started | 5088 | 5066
Completed | 4993 | 4976
Not Completed | 95 | 90
Not completed — Lost to Follow-up | 94 | 89
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Institutional review board request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Daily Vitamin Supplements: 1000mg of Vitamin C and 400IU of Vitamin E per capsule, twice daily between randomization (at 9 to 16 weeks) up to delivery.
- Placebo for Vitamins C and E: Placebo capsules consisting of Mineral Oil, Hydrogenated Vegetable Oil, Lecithin, Yellow wax, Soft Gelatin Shell, twice daily between randomization (at 9 to 16 weks) up to delivery.
- Total: Total of all reporting groups
Arm/Group | Daily Vitamin Supplements | Placebo for Vitamins C and E | Total
Number analyzed (Participants) | 5087 | 5065 | 10152
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (5.2) | 23.5 (5.2) | 23.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5087 | 5065 | 10152
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race or ethnic group was self-reported.
  Participants
    Black | 1268 | 1295 | 2563
    Hispanic | 1602 | 1566 | 3168
    Other | 2217 | 2204 | 4421
Week of pregnancy at randomization [Mean (Standard Deviation); unit: weeks] | 13.4 (2.1) | 13.4 (2.1) | 13.4 (2.1)
<13th week of pregnancy at randomization [Count of Participants; unit: Participants] | 2227 | 2203 | 4430
Prepregnancy body-mass index [Mean (Standard Deviation); unit: kg/m2] — The body-mass index is the weight in kilograms divided by the square of the height in meters. Prepregnancy weight used to calculate body-mass index was self-reported. Values were unavailable for 99 women in the vitamin group and 111 in the placebo group.
  kg/m2 | 25.4 (6.0) | 25.4 (5.9) | 25.4 (6.0)
Smoker [Count of Participants; unit: Participants] | 812 | 781 | 1593
Educational level [Mean (Standard Deviation); unit: year] | 12.8 (2.7) | 12.8 (2.7) | 12.8 (2.7)
Use of prenatal vitamins or multivitamins [Count of Participants; unit: Participants] | 3903 | 3889 | 7792
Daily dose of vitamin C [Median (Inter-Quartile Range); unit: mg] | 120 [50 to 120] | 100 [50 to 120] | 100 [50 to 120]
Daily dose of vitamin E [Median (Inter-Quartile Range); unit: IU] | 22 [3 to 30] | 22 [0 to 30] | 22 [2 to 30]
Previous pregnancy [Count of Participants; unit: Participants] | 1161 | 1170 | 2331
Family history of preeclampsia [Count of Participants; unit: Participants] — Family history is based on self-reported preeclampsia in a first-degree relative (mother, sister, or grandmother).
  Participants | 650 | 674 | 1324
Blood pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic | 109 (10) | 109 (10) | 109 (9.1)
  Diastolic | 66 (8) | 65 (8) | 65 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Composite of Pregnancy-associated Hypertension and Serious Adverse Outcomes in the Mother or Fetus or Neonate
Description: Severe hypertension (blood pressure [BP]>= 160/110) or mild hypertension (BP>= 140/90) >= 20 weeks gestation in conjunction with one of the following: elevated liver enzymes, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, an indicated preterm birth before 32 weeks of gestation owing to hypertension-related disorders, a fetus that was small for gestational age (below 3rd percentile) adjusted for sex and race or ethnic group, fetal death after 20 weeks of gestation, or neonatal death
Time Frame: 20 weeks through discharge following delivery
Population: The analysis was intent to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 305 | 285
Statistical Analysis 1: Comparison: Vitamins vs Placebo; The primary hypothesis states that antioxidant therapy initiated prior to 16 weeks gestation in women will reduce the frequency of serious maternal and infant complications associated with pregnancy related hypertension. We estimated that with a sample size of 10,000 women, the study would have 90% power to show a 30% reduction in the rate of the primary outcome, from 4% in the placebo to 2.8% in the vitamin group, with a two-sided type I error rate of 5%; Test type: Superiority or Other; p = 0.42, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.91 to 1.25]

2. Primary Outcome: Severe Hypertension
Description: Included here are women who had severe hypertension only and those who had severe hypertension with elevated liver enzyme levels, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, medically indicated preterm birth, fetal-growth restriction, or fetal death after 20 weeks of gestation, or neonatal death.
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 210 | 204
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.79, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.85 to 1.24]

3. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With Elevated Liver Enzyme Levels
Description: Elevated liver enzyme levels are specified as an aspartate aminotransferase level of >= 100 U per liter. Women who met more than one component of the primary outcome were counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 26 | 33
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.35, Chi-squared; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.47 to 1.31]

4. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With Thrombocytopenia
Description: Thrombocytopenia defined as a platelet count of <100,000 per cubic millimeter. Women who met more than one component of the primary outcome were counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Time Frame: 20 weeks through discharge following delivery
Measure: Number; unit: participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
participants | 21 | 31
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.16, Chi-squared; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.39 to 1.17]

5. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With an Elevated Serum Creatinine Level
Description: Elevated serum creatinine defined as ≥1.5 mg per deciliter or 132.6 μmol per liter. Women who met more than one component of the primary outcome were counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 7 | 11
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.34, Chi-squared; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.25 to 1.63]

6. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With an Eclamptic Seizure
Description: Women who met more than one component of the primary outcome were counted for each component. Therefore, the number of women for all individual components combined is greater than the number of women with the primary outcome.
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 10 | 4
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.11, Chi-squared; Risk Ratio (RR) = 2.49, 95% CI 2-sided [0.78 to 7.94]

7. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With an Indicated Preterm Birth Before 32 Weeks of Gestation Owing to Hypertension-related Disorders
Description: as for outcome 6
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 13 | 16
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.57, Chi-squared; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.39 to 1.68]

8. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With a Fetus That Was Small for Gestational Age (Below the 3rd Percentile) Adjusted for Sex and Race or Ethnic Group
Description: as for outcome 6
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 60 | 46
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.18, Chi-squared; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.89 to 1.90]

9. Primary Outcome: Severe or Mild Pregnancy-associated Hypertension With a Fetal Death After 20 Weeks of Gestation or Neonatal Death
Description: as for outcome 6
Time Frame: 20 weeks through discharge or prior to discharge following delivery admission
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 12 | 11
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.84, Chi-squared; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.48 to 2.46]

10. Secondary Outcome: Preeclampsia (Mild, Severe, HELLP Syndrome, Eclampsia)
Description: HELLP denotes hemolytic anemia, elevated liver enzymes, and low platelet count.
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants
  Total Preeclampsia | 358 | 332
  Mild Preeclampsia | 212 | 191
  Severe Preeclampsia | 134 | 129
  HELLP Syndrome | 2 | 8
  Eclampsia | 10 | 4
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.33, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.93 to 1.24]

11. Secondary Outcome: Pregnancy Associated Hypertension
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 1457 | 1322
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.004, Chi-squared; Risk Ratio (RR) = 1.10, 95% CI 2-sided [1.03 to 1.17]

12. Secondary Outcome: Medically Indicated Delivery Because of Hypertension
Time Frame: 20 weeks through discharge following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4952 | 4934
Participants | 509 | 473
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.25, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.95 to 1.21]

13. Secondary Outcome: Aspartate Aminotransferase ≥100 U/Liter
Time Frame: 20 weeks through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 35 | 48
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.15, Chi-squared; Risk Ratio (RR) = 0.73, 95% CI [0.47 to 1.12]

14. Secondary Outcome: Creatinine ≥1.5 mg/dl (133 μmol/Liter)
Time Frame: 20 weeks through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants | 9 | 12
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.51, Chi-squared; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.32 to 1.77]

15. Secondary Outcome: Antepartum Bleeding
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4956 | 4937
Participants | 56 | 46
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.33, Chi-squared; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.82 to 1.79]

16. Secondary Outcome: Premature Rupture of Membranes
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4934 | 4923
Participants | 124 | 129
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.74, Chi-squared; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.75 to 1.22]

17. Secondary Outcome: Placental Abruption
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4957 | 4938
Participants | 24 | 36
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.12, Chi-squared; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.40 to 1.11]

18. Secondary Outcome: Cesarean Delivery
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4958 | 4940
Participants | 1269 | 1224
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.35, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.97 to 1.11]

19. Secondary Outcome: Maternal Death
Time Frame: Delivery through hospital discharge
Population: One maternal death in each group due to peripartum cardiomyopathy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dietary Supplement/Vitamins | Placebo for Vitamin C and Vitamin E
Number analyzed (Participants) | 4993 | 4976
Participants | 1 | 1

20. Secondary Outcome: Postpartum Pulmonary Edema
Time Frame: After delivery through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4951 | 4926
Participants | 3 | 10
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.30, 95% CI 2-sided [0.08 to 1.08]

21. Secondary Outcome: Hematocrit ≤24% With Transfusion
Time Frame: Delivery admission to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4954 | 4927
Participants | 40 | 59
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.45 to 1.01]

22. Secondary Outcome: Maternal Hospital Stay
Time Frame: Delivery through discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4952 | 4935
days | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Gestational Age at Delivery
Time Frame: Delivery
Measure: Median (Standard Deviation); unit: weeks
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
weeks | 38.9 (3.5) | 38.8 (3.5)
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Preterm Birth
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants
  <37 weeks' gestation | 513 | 526
  <32 weeks' gestation | 149 | 173
Statistical Analysis 1: Comparison: Vitamins vs Placebo; <37 weeks' gestation; Test type: Superiority or Other; p = 0.63, Chi-squared; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.87 to 1.09]
Statistical Analysis 2: Comparison: Vitamins vs Placebo; <32 weeks' gestation; Test type: Superiority or Other; p = 0.16, Chi-squared; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.69 to 1.06]

25. Secondary Outcome: Fetal or Neonatal Death
Time Frame: During pregnancy or thorugh discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4993 | 4976
Participants
  All Fetal or Neonatal Deaths | 113 | 122
  Fetal loss at < 20 weeks | 55 | 59
  Fetal death at ≥20 weeks | 38 | 36
  Neonatal death | 20 | 27
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.53, Chi-squared; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.72 to 1.19]

26. Secondary Outcome: Birth Weight
Time Frame: At birth
Population: Liveborn infants
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
grams | 3247 (575) | 3244 (581)
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Small for Gestational Age
Description: A baby whose birth weight is less than the 3rd percentile is considered to be small for gestational age (adjusted for sex and race or ethnic group)
Time Frame: At birth
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 133 | 132
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.98, Chi-squared; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.79 to 1.27]

28. Secondary Outcome: Birth Weight <2500 Grams
Time Frame: At birth
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 345 | 369
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.32, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.81 to 1.07]

29. Secondary Outcome: Admission to NICU
Description: NICU denotes neonatal intensive care unit.
Time Frame: Delivery through discharge
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 577 | 557
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.58, Chi-squared; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.92 to 1.15]

30. Secondary Outcome: Respiratory Distress Syndrome
Time Frame: Delivery through discharge
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 150 | 144
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.75, Chi-squared; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.83 to 1.30]

31. Secondary Outcome: Intraventricular Hemorrhage, Grade III or IV
Time Frame: Delivery through discharge
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 6 | 7
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.78, Chi-squared; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.29 to 2.54]

32. Secondary Outcome: Sepsis
Time Frame: Delivery through discharge
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 30 | 23
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.34, Chi-squared; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.76 to 2.23]

33. Secondary Outcome: Necrotizing Enterocolitis
Time Frame: Delivery through discharge
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 10 | 14
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.41, Chi-squared; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.32 to 1.60]

34. Secondary Outcome: Retinopathy of Prematurity
Time Frame: Within 1 month of birth
Population: Live born infants
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
Participants | 19 | 16
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.62, Chi-squared; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.61 to 2.30]

35. Secondary Outcome: Apgar Score <=3 at 5 Minutes
Time Frame: At birth
Measure: Number; unit: participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
participants | 23 | 27
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.56, Chi-squared; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.49 to 1.48]

36. Secondary Outcome: Neonatal Hospital Stay
Time Frame: Birth through discharge from hospital
Population: Live born infants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 4900 | 4881
days | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

37. Post Hoc Outcome: Analysis of Primary Composite Outcome in Participants Randomized on or After the 13th Week of Pregnancy
Description: Subgroup analysis of the primary composite outcome (severe pregnancy associated hypertension or severe or mild hypertension with elevated liver-enzyme levels, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, indicated preterm birth, fetal-growth restriction or prenatal death) in participants who were randomized on or after the 13th week of pregnancy.
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Vitamins: 1000mg of Vitamin C and 400IU of Vitamin E per capsule, twice daily between randomization (at 9 to 16 weeks) up to delivery.
  Dietary Supplement/Vitamins: Vitamin C (1000 mg) and Vitamin E (400 IU) per capsule, two capsules daily between randomization (at 9 - 16 weeks gestation) up to delivery.
- Placebo: Placebo capsules consisting of Mineral Oil, Hydrogenated Vegetable Oil, Lecithin, Yellow wax, Soft Gelatin Shell, twice daily between randomization (at 9 to 16 weks) up to delivery.
  Placebo for Vitamin C and Vitamin E: Placebo two capsules daily between randomization (at 9 - 16 weeks gestation) up to delivery.
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 2812 | 2814
Participants | 161 | 158
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.86, Chi-squared; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.82 to 1.26]

38. Post Hoc Outcome: Analysis of Primary Composite Outcome in Participants Randomized Before the 13th Week of Pregnancy
Description: Subgroup analysis of the primary composite outcome (severe pregnancy associated hypertension or severe or mild hypertension with elevated liver-enzyme levels, thrombocytopenia, elevated serum creatinine levels, eclamptic seizure, indicated preterm birth, fetal-growth restriction or prenatal death) in participants who were randomized before the 13th week of pregnancy.
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamins | Placebo
Number analyzed (Participants) | 2181 | 2162
Participants | 144 | 127
Statistical Analysis 1: Comparison: Vitamins vs Placebo; Test type: Superiority or Other; p = 0.32, Chi-squared; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.89 to 1.42]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning with enrollment (between 9 weeks 0 days gestation and 16 weeks 6 days gestation) through the duration of the pregnancy, delivery, and hospital discharge for the mother and baby. This time period varies by participant and may cover anywhere from 9 weeks gestation to 42 weeks gestation.
Arm/Group | Vitamins | Placebo
All-Cause Mortality (participants affected / at risk) | 1/5087 | 1/5065
Serious Adverse Events (participants affected / at risk) | 108/5087 | 173/5065
Other Adverse Events (participants affected / at risk) | 0/5087 | 0/5065
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamins (N=5087) | Placebo (N=5065)
Peripartum Cardiomyopathy (Cardiac disorders) | 1 | 1 — Peripartum Cardiomyopathy resulting in death.
Fetal Death (Pregnancy, puerperium and perinatal conditions) | 45 | 95 — Miscarriage, stillbirth, abortion
Bleeding (Pregnancy, puerperium and perinatal conditions) | 9 | 7 — Placental abruption, vaginal bleeding
Renal and Urinary disorders (Renal and urinary disorders) | 4 | 9 — Pyelonephritis and Urinary Tract Infection
Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 4 | 5 — Postpartum hemorrhage, blood transfusion, hysterectomy
Infection (Infections and infestations) | 5 | 2 — Group A strep sepsis, bacterial/ viral meningitis, cellulitis, sepsis, bacterial infection
Respiratory distress/pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DVT/PE (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — Deep vein thrombosis, pulmonary embolism
Colon resection (Surgical and medical procedures) | 1 | 0
Hodgkin's disease (Blood and lymphatic system disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Fetal birth defects (Congenital, familial and genetic disorders) | 6 | 21
Fetal atrial flutter/arrythmia/bradycardia (Congenital, familial and genetic disorders) | 2 | 1
Neonatal death (General disorders) | 20 | 27
Infant Seizures (Nervous system disorders) | 2 | 0
Birth injury (Injury, poisoning and procedural complications) | 1 | 1
Infant low platelet count (Blood and lymphatic system disorders) | 1 | 0
Infant - Soft Tissue Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Umbilical hernia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoxic Events (Nervous system disorders) | 2 | 0 — Hypoxic birth injury, hypoxic ischemic encephalopathy, ischemic stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less